CLINICAL TRIAL: NCT00694161
Title: The Effects Of Fx-1006A On Transthyretin Stabilization And Clinical Outcome Measures In Patients With V122I Or Wild-Type TTR Amyloid Cardiomyopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FX1B-201; B3461025
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Results first posted 2012-12-18 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Cardiomyopathy
Keywords: Transthyretin; TTR; ATTR; TTR amyloidosis; cardiomyopathy; V122I; wild-type TTR; SSA; Patients with V122I or wild-type TTR amyloid cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies | interventions — tafamidis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fx-1006A (Experimental)
  Interventions: Drug: Fx-1006A

INTERVENTIONS:
Drug: Fx-1006A — Fx-1006A 20mg soft gelatin capsules once daily (at the same time each day) for 12 months

SUMMARY:
Open-label, multicenter, international, single-treatment study designed to determine TTR stabilization as well as Fx-1006A safety and tolerability, and its effects on clinical outcomes in patients with V122I or wild-type TTR amyloid cardiomyopathy.

The study will be conducted in two parts. Part 1 will include a six-week dosing period during which all enrolled patients will self-administer oral Fx-1006A 20 mg soft gelatin capsules once daily for six weeks. At Week 6, blood samples will be collected from each patient to determine TTR stabilization. Patients who complete the Week 6 visit will continue taking daily oral Fx 1006A 20 mg for up to a total of 12 months during Part 2 of this study. If it is determined that a patient is not stabilized at Week 6 (based on TTR stabilization data), the patient will be discontinued from the study. Safety and clinical outcomes will be evaluated during Part 2 of this study.

Two whole blood samples for pharmacodynamic assessments (TTR stabilization) and pharmacokinetic assessments (Fx-1006A concentrations as well as calculated steady-state parameters) will be collected at Baseline and Week 6. At Months 6 and 12, two whole blood samples will be collected for pharmacodynamic assessments, and four whole blood samples (two samples per time point) will be collected for pharmacokinetic assessments to be utilized in population pharmacokinetic modeling.

Echocardiography, chest x-ray, cardiac MRI, and 24-hour Holter monitoring will be conducted at Baseline, and Months 6 and 12. Six-minute walk test and quality of life utilizing the Patient Global Assessment, KCCQ, and SF-36 will be assessed at Baseline, and Months 3, 6, and 12. NYHA Classification will be assessed at Baseline, Week 6, and Months 3, 6, and 12. Serum markers of troponin I and T, and NT-pro-BNP levels will be assessed at each study visit.

Safety and tolerability will be assessed throughout the study. Vital signs, 12-lead ECG, blood and urine samples for clinical laboratory tests (serum chemistry, hematology, coagulation panel, and urinalysis), AEs, and concomitant medications (including diuretic usage) will be assessed at each study visit. Abbreviated physical examinations will be conducted at Baseline, Weeks 2 and 6, and Months 3 and 6, and a complete physical examination will be conducted at Month 12.

Clinic visits will be conducted during Screening (Days -30 to -1) and Baseline (Day 0); procedures scheduled for the Baseline visit may be conducted over a period of one week to accommodate patient scheduling. All Baseline procedures must be completed prior to the first self-administered dose on Day 1. Day 1 will be defined as administration of the first dose of study medication, which patients will self-administer at home. During treatment, clinic visits will be conducted at Week 2 (± 2 days), Week 6 (± 1 week), Month 3 (± 1 week), Month 6 (± 2 weeks), and Month 12 (± 2 weeks). Procedures scheduled for the Month 6 and 12 visits may occur over one week during the visit window to accommodate patient scheduling. Monthly telephone contacts (± 1 week of the scheduled date) will be made during months in which no clinical site visits are scheduled (Months 4, 5, 7, 8, 9, 10, and 11) for assessment of AEs and concomitant medications. A final telephone contact to assess AEs and concomitant medication usage will be made 30 days after the last dose of study medication for each patient.

Patients who discontinue from the study at any time will have a final visit performed, including all safety assessments, at the time of discontinuation. Any patient discontinuing after the Month 6 visit will also have all exploratory assessments performed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is > 40 years-old.
2. Patient participated in FoldRx Study Fx-001 (TRACS) OR Patient has documented TTR amyloid cardiomyopathy and NYHA Classification of I or II.

   TTR amyloid cardiomyopathy is defined as:
   1. Variant TTR amyloid cardiomyopathy as defined as: V122I genotype and presence of amyloid in cardiac biopsy tissue (as determined by congo red stain, alcin blue stain, or immunohistochemical TTR analysis), or
   2. Variant TTR amyloid cardiomyopathy as defined as: V122I genotype, evidence of cardiac involvement by echocardiography with left ventricle wall thickness > 12 mm and presence of amyloid in non-cardiac biopsy tissue (as determined by congo red stain, alcin blue stain, or immunohistochemical TTR analysis), or
   3. Wild-type TTR amyloid cardiomyopathy as defined as: normal TTR genotype and presence of TTR amyloid deposits in cardiac biopsy tissue (as determined by congo red stain and immunohistochemical TTR analysis), or
   4. Wild-type TTR amyloid cardiomyopathy as defined as: normal TTR genotype, evidence of cardiac involvement by echocardiography with left ventricle wall thickness > 12 mm and presence of TTR amyloid deposits in non-cardiac biopsy tissue (as determined by congo red stain and immunohistochemical TTR analysis).
3. Patient's symptoms of congestive heart failure (CHF) have been optimally managed prior to baseline, as assessed by the Principal Investigator. Optimal CHF management includes stable drug regimen for ≥ 4 weeks prior to enrollment and stable dose of beta blocker for ≥ 3 months prior to enrollment.
4. If female, patient is post-menopausal. If male with a female partner of childbearing potential, willing to use an acceptable method of birth control for the duration of the study and for at least 3 months after the last dose of study medication.
5. Patient is, in the opinion of the Investigator, willing and able to comply with the study medication regimen and all other study requirements

Exclusion Criteria:

1. Chronic use of non-protocol approved non-steroidal anti-inflammatory drugs (NSAIDs), defined as greater than 3-4 times/month. The following NSAID are allowed: acetylsalicylic acid, etodolac, ibuprofen, indomethicin, ketoprofen, nabumetone, naproxen, nimesulide, piroxicam, and sulindac.
2. Patient has a TTR mutation other than V122I.
3. Patient has primary or secondary amyloidosis.
4. Patient has received prior liver or heart transplantation.
5. Patient with positive results for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (anti-HCV), and/or human immunodeficiency virus (HIV).
6. Patient has renal failure requiring dialysis.
7. Patient has moderate or severe hepatic impairment (assessed by Child-Pugh).
8. Patient has liver function test abnormalities: alanine transaminases (ALT) and/or aspartate transaminases (AST) > 2 times upper limit of normal (ULN) that, in the medical judgment of the Investigator, are due to reduced liver function or active liver disease.
9. Patient has prior non-amyloid cardiac disease, such as myocardial infarction due to obstructive coronary artery disease, active non-amyloid cardiomyopathy (i.e., symptomatic left ventricular dysfunction from any cause other than amyloid), or symptomatic valvular heart disease that significantly contribute to the patient's underlying cardiac signs or symptoms.
10. Patient has a co-morbidity anticipated to limit survival to less than 12 months.
11. Patient received an investigational drug/device in another clinical investigational study within 60 days before Baseline (Day 0).
12. Patient had active alcohol or substance abuse within 60 days before Baseline (Day 0).
13. Patient has a history of documented noncompliance.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Packman, MBA, Study Director — FoldRx Pharmaceuticals, Inc
Locations (6):
- United States (6):
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Harvard Vanguard Medical Associates, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University, New York, New York

REFERENCES:
- [Derived] Sultan MB, Gundapaneni B, Schumacher J, Schwartz JH. Treatment With Tafamidis Slows Disease Progression in Early-Stage Transthyretin Cardiomyopathy. Clin Med Insights Cardiol. 2017 Sep 18;11:1179546817730322. doi: 10.1177/1179546817730322. eCollection 2017. PMID 28951660
- [Derived] Maurer MS, Grogan DR, Judge DP, Mundayat R, Packman J, Lombardo I, Quyyumi AA, Aarts J, Falk RH. Tafamidis in transthyretin amyloid cardiomyopathy: effects on transthyretin stabilization and clinical outcomes. Circ Heart Fail. 2015 May;8(3):519-26. doi: 10.1161/CIRCHEARTFAILURE.113.000890. Epub 2015 Apr 14. PMID 25872787

RESULTS

PARTICIPANT FLOW:
Groups:
- Tafamidis: Participants with variant transthyretin (TTR) genotype (valine replaced at position 122 by isoleucine or V122I) and wild-type TTR genotype received tafamidis (Fx-1006A) 20 milligram (mg) capsule orally once daily up to Week 6 in Part 1 and participants who achieved TTR stabilization at Week 6 continued to receive tafamidis (Fx-1006A) 20 mg capsule orally once daily up to Month 12 in Part 2.
Period: Part 1 (up to Week 6)
Arm/Group | Tafamidis
Started | 35
Completed | 35
Not Completed | 0
Period: Part 2 (After Week 6 up to Month 12)
Arm/Group | Tafamidis
Started | 35
Completed | 32
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tafamidis
Number analyzed (Participants) | 35
Age Continuous [Mean (Standard Deviation); unit: Years] | 76.4 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 32

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Stabilized Transthyretin (TTR Tetramer) at Week 6
Description: TTR tetramer was assessed using a validated immunoturbidimetric assay. The Fraction of Initial (FOI) is the ratio of the measured TTR tetramer concentration after denaturation to the measured TTR tetramer concentration before denaturation. TTR tetramer stabilization is based on the difference between the on-treatment FOI and the baseline FOI expressed as a percentage of the baseline FOI.
Time Frame: Week 6
Population: Intent-to-Treat (ITT) population included all participants who received at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tafamidis
Number analyzed (Participants) | 35
Percentage of participants | 97.1 [85.1 to 99.9]

2. Secondary Outcome: Percentage of Participants With Stabilized Transthyretin (TTR Tetramer) at Month 6 and 12
Description: as for outcome 1
Time Frame: Month 6, Month 12
Population: ITT population included all participants who received at least one dose of study medication. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tafamidis
Number analyzed (Participants) | 34
Percentage of participants
  Month 6 | 88.2 [72.5 to 96.7]
  Month 12 | 87.5 [71.0 to 96.5]

3. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent are events between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 30 days after the last dose
Population: ITT population included all participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Tafamidis
Number analyzed (Participants) | 35
Participants | 35

4. Other Pre Specified Outcome: Number of Participants With Greater Than or Equal to (>=) Grade 3 Treatment-Emergent AEs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent are events between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state. On the basis of intensity, grade 3 was referred as severe, grade 4 as life-threatening and grade 5 as death.
Time Frame: Baseline up to 30 days after the last dose
Population: ITT population included all participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Tafamidis
Number analyzed (Participants) | 35
Participants
  Grade 3 (severe) | 18
  Grade 4 (life-threatening) | 1
  Grade 5 (death) | 2

5. Other Pre Specified Outcome: Number of Participants With Clinically Significant Treatment-Emergent Echocardiography (ECHO) Findings
Description: ECHO:investigator assessed test to assess cardiac function.ECHO abnormality criteria:any/valvular abnormality,pericardial effusion,abnormal regional wall motion,inferior vena cava respiratory variation,posterior left ventricular wall/septal thickness>=13 millimeter(mm),right ventricular thickness>=7mm,ejection fraction <50%, ratio of early (E) diastolic transmitral flow and atrial(A) contraction velocity (E/A)>=2, ratio of 'E'to lateral/septal mitral annular velocity (e') (E/e'prime lateral>15, E/e'prime septal>15), E deceleration time<=150 millisecond(msec),Isovolumic relaxation time<=70msec.
Time Frame: Baseline up to Month 12
Population: ITT population. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. The 'n' for any post-dose incidence included participants with baseline values that were not abnormal(that is treatment-emergent abnormalities).
Measure: Number; unit: Participants
Arm/Group | Tafamidis
Number analyzed (Participants) | 34
Participants
  Any ECHO abnormalities (n=34) | 31
  Pericardial effusion (n=28) | 6
  Valvular abnormalities- thickening (n=4) | 4
  Valvular abnormalities- regurgitation (n=7) | 6
  Abnormal regional wall motion (n=19) | 10
  Inferior vena cava respiratory variation (n=14) | 7
  Left ventricular posterior wall thickness (n=0) | NA — Data not analyzed since no participant were eligible for analysis.
  Left ventricular septal thickness (n=0) | NA — Data not analyzed since no participant were eligible for analysis.
  Right ventricular thickness (n=7) | 6
  E/A ratio (n=8) | 4
  E/e' prime lateral (n=13) | 5
  E/e' prime septal (n=6) | 5
  Ejection fraction (n=18) | 11
  E deceleration time (n=16) | 8
  Isovolumic relaxation time (n=16) | 4

6. Other Pre Specified Outcome: Number of Participants Discontinuing From The Study Due to Clinically Significant Clinical or Laboratory Adverse Events (AEs)
Time Frame: Baseline up to Month 12
Population: ITT population included all participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Tafamidis
Number analyzed (Participants) | 35
Participants | 1

7. Other Pre Specified Outcome: Change From Baseline in Echocardiographic (ECHO) Parameters at Month 6 and 12
Description: Echocardiography was used to measure interventricular septal thickness (IVST), posterior left ventricular wall thickness (PLVWT), right ventricular wall thickness (RVWT), left atrial diameter (LAD): anterior-posterior (ant-post), medio-lateral, superior-inferior (sup-inf) and left ventricular end diastolic diameter (LVEDD).
Time Frame: Baseline, Month 6, Month 12
Population: ITT population included all participants who received at least one dose of study medication. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. Here 'n' signifies those participants who were evaluable for specific timepoints.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Tafamidis
Number analyzed (Participants) | 34
millimeter (mm)
  IVST: Baseline (n=34) | 20.71 (3.58)
  IVST: Change at Month 6 (n=33) | -0.64 (2.41)
  IVST: Change at Month 12 (n=30) | 0.87 (2.52)
  PLVWT: Baseline (n=34) | 20.20 (3.37)
  PLVWT: Change at Month 6 (n=33) | -0.50 (3.83)
  PLVWT: Change at Month 12 (n=30) | -0.00 (2.11)
  RVWT: Baseline (n=27) | 9.21 (2.34)
  RVWT: Change at Month 6 (n=21) | -0.47 (2.47)
  RVWT: Change at Month 12 (n=20) | 0.26 (2.25)
  LAD (ant-post): Baseline (n=34) | 45.00 (6.14)
  LAD (ant-post): Change at Month 6 (n=33) | -0.40 (4.33)
  LAD (ant-post): Change at Month 12 (n=30) | -0.30 (4.19)
  LAD (medio-lateral): Baseline (n=34) | 44.10 (5.56)
  LAD (medio-lateral): Change at Month 6 (n=32) | 0.70 (5.17)
  LAD (medio-lateral): Change at Month 12 (n=30) | -0.90 (6.41)
  LAD (sup-inf): Baseline (n=34) | 61.50 (8.43)
  LAD (sup-inf): Change at Month 6 (n=32) | 3.00 (5.90)
  LAD (sup-inf): Change at Month 12 (n=30) | 0.80 (6.29)
  LVEDD: Baseline (n=34) | 37.94 (5.19)
  LVEDD: Change at Month 6 (n=33) | 0.45 (3.49)
  LVEDD: Change at Month 12 (n=30) | 0.10 (3.41)

8. Other Pre Specified Outcome: Change From Baseline in Left Ventricular Mass (LVM) at Month 6 and 12
Description: LVM was defined as increase in the mass of left ventricle, estimated by echocardiography. Increased LVM was associated with cardiovascular morbidity and mortality.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Gram
Arm/Group | Tafamidis
Number analyzed (Participants) | 34
Gram
  Baseline (n=34) | 372.50 (123.96)
  Change at Month 6 (n=33) | -19.76 (54.38)
  Change at Month 12 (n=30) | 13.73 (77.12)

9. Other Pre Specified Outcome: Change From Baseline in Left Ventricular Ejection Fraction at Month 6 and 12
Description: Left ventricular ejection fraction (LVEF) was the fraction of the end-diastolic volume (EDV) that is ejected out of left ventricle with each contraction, estimated by echocardiography. EDV is the volume of blood within a ventricle immediately before a contraction.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage of EDV
Arm/Group | Tafamidis
Number analyzed (Participants) | 34
Percentage of EDV
  Baseline (n=34) | 46.8 (14.1)
  Change at Month 6 (n=33) | -0.4 (10.3)
  Change at Month 12 (n=30) | -3.7 (10.4)

10. Other Pre Specified Outcome: Change From Baseline in Doppler Data: E/A and E/e' Ratio at Month 6 and 12
Description: Doppler echocardiography was a procedure which used ultrasound technology to examine the heart. Ratio of early (E) diastolic transmitral flow velocity and atrial (A) contraction velocity (E/A) and ratio of the early (E) diastolic transmitral flow velocity to the mitral annular velocity (e') (E/e') were estimated.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Tafamidis
Number analyzed (Participants) | 26
Ratio
  E/A ratio: Baseline (n=19) | 2.516 (1.084)
  E/A ratio: Change at Month 6 (n=12) | 0.425 (1.117)
  E/A ratio: Change at Month 12 (n=9) | 0.544 (0.575)
  E/e' ratio: Baseline (n=26) | 16.240 (9.089)
  E/e' ratio: Change at Month 6 (n=15) | 2.217 (3.166)
  E/e' ratio: Change at Month 12 (n=14) | -0.717 (5.681)

11. Other Pre Specified Outcome: Change From Baseline in Doppler Data: Mitral Deceleration Time at Month 6 and 12
Description: Doppler echocardiography was a procedure which used ultrasound technology to examine the heart. The mitral deceleration time was the time taken from the maximum E wave to baseline. E wave arises due to early diastolic filling.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Tafamidis
Number analyzed (Participants) | 33
msec
  Baseline (n=33) | 152.9 (35.3)
  Change at Month 6 (n=27) | 1.0 (37.5)
  Change at Month 12 (n=27) | -7.1 (32.6)

12. Other Pre Specified Outcome: Change From Baseline in Tissue Doppler- Septal and Lateral Velocity at Month 6 and 12
Description: Tissue Doppler used doppler principles to measure the annular velocities at the lateral and septal areas of the mitral annulus. s': systolic velocity during ejection, e': early diastolic mitral annular velocity, a': late diastolic mitral annular velocity.
Time Frame: Baseline, Month 6, Month 12
Population: ITT population included all participants who received at least one dose of study medication. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. Here 'n' signifies those participants who were evaluable for specific categories.
Measure: Mean (Standard Deviation); unit: centimeter/second (cm/sec)
Arm/Group | Tafamidis
Number analyzed (Participants) | 26
centimeter/second (cm/sec)
  Septal s': Baseline (n=23) | 3.70 (1.31)
  Septal s': Change at Month 6 (n=16) | -0.57 (0.73)
  Septal s': Change at Month 12 (n=14) | -0.69 (0.77)
  Septal e': Baseline (n=23) | 3.67 (1.60)
  Septal e': Change at Month 6 (n=17) | -0.09 (1.12)
  Septal e': Change at Month 12 (n=14) | -0.33 (1.32)
  Septal a': Baseline (n=16) | 2.51 (1.60)
  Septal a': Change at Month 6 (n=6) | -0.40 (0.43)
  Septal a': Change at Month 12 (n=6) | -0.42 (0.72)
  Lateral s': Baseline (n=24) | 4.53 (1.59)
  Lateral s': Change at Month 6 (n=14) | -0.50 (1.16)
  Lateral s': Change at Month 12 (n=13) | -0.73 (1.22)
  Lateral e': Baseline (n=26) | 5.09 (2.00)
  Lateral e': Change at Month 6 (n=16) | -0.76 (0.80)
  Lateral e': Change at Month 12 (n=14) | 0.05 (0.88)
  Lateral a': Baseline (n=17) | 3.16 (1.94)
  Lateral a': Change at Month 6 (n=7) | -0.41 (0.60)
  Lateral a': Change at Month 12 (n=9) | 0.06 (1.03)

13. Other Pre Specified Outcome: Change From Baseline in Pericardial Effusion at Month 6 and 12
Description: Pericardial effusion was the presence of an abnormal amount of fluid in the pericardial cavity, as determined by echocardiography.
Time Frame: Baseline, Month 6, Month 12
Population: Data for this pre-specified outcome measure was collected and reported in individual participant listings but not statistically summarized for analysis.
Arm/Group | Tafamidis
Number analyzed (Participants) | 0

14. Other Pre Specified Outcome: Number of Participants With Change From Baseline in Valvular Abnormalities at Month 6 and 12
Description: Valvular abnormalities were those abnormalities (thickening or regurgitation) that involved one or more valves of the heart, determined by echocardiography.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 13
Arm/Group | Tafamidis
Number analyzed (Participants) | 0

15. Other Pre Specified Outcome: Change From Baseline in Left Ventricular Anteroseptal, Left Ventricular Inferolateral Wall Thickness and Right Ventricular End Diastolic Free Wall Thickness at Month 6 and 12
Description: Cardiac Magnetic Resonance Imaging (MRI) was done to measure the thickness of left ventricular anteroseptal (LVAS) wall, left ventricular inferolateral (LVIL) wall and right ventricular end diastolic free (RVEDF) wall.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tafamidis
Number analyzed (Participants) | 18
mm
  LVAS wall thickness: Baseline (n=18) | 15.808 (3.603)
  LVAS wall thickness: Change at Month 6 (n=18) | 0.810 (3.447)
  LVAS wall thickness: Change at Month 12 (n=15) | 0.813 (3.099)
  LVIL wall thickness: Baseline (n=18) | 15.405 (4.616)
  LVIL wall thickness: Change at Month 6 (n=18) | -1.472 (4.333)
  LVIL wall thickness: Change at Month 12 (n=15) | 1.182 (4.782)
  RVEDF wall thickness: Baseline (n=17) | 10.871 (14.001)
  RVEDF wall thickness: Change at Month 6 (n=17) | -4.501 (14.734)
  RVEDF wall thickness: Change at Month 12 (n=15) | -1.577 (4.722)

16. Other Pre Specified Outcome: Change From Baseline in Left Ventricular Mass, Mass of Left Ventricular Myocardium With Amyloidosis, Mass of Left Ventricular Myocardium With Fibrosis/Scar and Right Ventricular End Diastolic Mass at Month 6 and 12
Description: Cardiac MRI was done to measure LVM, mass of left ventricular (LV) myocardium with amyloidosis, mass of LV myocardium with fibrosis/scar and right ventricular end diastolic mass (RVEDM).
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Gram
Arm/Group | Tafamidis
Number analyzed (Participants) | 18
Gram
  LVM: Baseline (n=18) | 221.599 (63.680)
  LVM: Change at Month 6 (n=18) | 0.557 (24.901)
  LVM: Change at Month 12 (n=15) | 0.119 (20.027)
  LV Amyloidosis: Baseline (n=15) | 63.963 (25.614)
  LV Amyloidosis : Change at Month 6 (n=14) | -13.854 (23.921)
  LV Amyloidosis: Change at Month 12 (n=9) | -4.346 (38.364)
  LV Fibrosis/Scar: Baseline (n=15) | 87.746 (60.297)
  LV Fibrosis/Scar: Change at Month 6 (n=14) | -30.496 (52.176)
  LV Fibrosis/Scar: Change at Month 12 (n=9) | -20.238 (64.487)
  RVEDM: Baseline (n=18) | 65.999 (20.296)
  RVEDM: Change at Month 6 (n=18) | -4.377 (20.648)
  RVEDM: Change at Month 12 (n=15) | 0.215 (18.038)

17. Other Pre Specified Outcome: Change From Baseline in Left Ventricle End Diastolic Volume, Left Ventricle End Systolic Volume, Left Ventricle Stroke Volume, Right Ventricle End Diastolic Volume, Right Ventricle End Systolic Volume, Right Ventricle Stroke Volume at Month 6 and 12.
Description: Cardiac MRI was done to measure left ventricle end diastolic volume (LVEDV), left ventricle end systolic volume (LVESV), left ventricle stroke volume (LVSV), right ventricle end diastolic volume (RVEDV), right ventricle end systolic volume (RVESV) and right ventricle stroke volume (RVSV).
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Tafamidis
Number analyzed (Participants) | 18
mL
  LVEDV: Baseline (n=18) | 166.673 (40.417)
  LVEDV: Change at Month 6 (n=18) | -0.922 (21.164)
  LVEDV: Change at Month 12 (n=15) | -1.606 (20.323)
  LVESV: Baseline (n=18) | 84.651 (29.271)
  LVESV: Change at Month 6 (n=18) | 3.727 (20.963)
  LVESV: Change at Month 12 (n=15) | 6.479 (16.810)
  LVSV: Baseline (n=18) | 82.022 (19.866)
  LVSV: Change at Month 6 (n=18) | -4.651 (21.391)
  LVSV: Change at Month 12 (n=15) | -8.083 (15.614)
  RVEDV: Baseline (n=18) | 175.124 (67.977)
  RVEDV: Change at Month 6 (n=18) | -4.836 (37.879)
  RVEDV: Change at Month 12 (n=15) | 19.540 (39.413)
  RVESV: Baseline (n=18) | 104.662 (48.775)
  RVESV: Change at Month 6 (n=18) | -1.727 (21.438)
  RVESV: Change at Month 12 (n=15) | 26.250 (30.858)
  RVSV: Baseline (n=18) | 70.478 (26.364)
  RVSV: Change at Month 6 (n=18) | -3.125 (26.125)
  RVSV: Change at Month 12 (n=15) | -6.730 (33.975)

18. Other Pre Specified Outcome: Change From Baseline in Left Ventricular Ejection Fraction and Right Ventricular Ejection Fraction at Month 6 and 12
Description: Cardiac MRI was done to measure: left ventricular ejection fraction (LVEF) was the fraction of the EDV that is ejected out of left ventricle with each contraction and right ventricular ejection fraction (RVEF) was the fraction of the EDV that is ejected out of right ventricle with each contraction. EDV is the volume of blood within a ventricle immediately before a contraction.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage of EDV
Arm/Group | Tafamidis
Number analyzed (Participants) | 18
Percentage of EDV
  LVEF: Baseline (n=18) | 50.176 (9.183)
  LVEF: Change at Month 6 (n=18) | -2.713 (13.362)
  LVEF: Change at Month 12 (n=14) | -3.511 (9.063)
  RVEF: Baseline (n=18) | 42.323 (11.949)
  RVEF: Change at Month 6 (n=18) | -1.756 (10.381)
  RVEF: Change at Month 12 (n=15) | -7.381 (12.040)

19. Other Pre Specified Outcome: Change From Baseline in Left Ventricular Cardiac Output and Right Ventricular Cardiac Output at Month 6 and 12
Description: Cardiac MRI was done to measure cardiac output, which was the volume of blood being pumped by the heart, in particular by the left or right ventricle in the time interval of one minute.
Time Frame: Baseline, Month 6, Month 12
Population: MRI data was collected and reported for cardiac output through the measure of stroke volume as given in outcome measure 17.
Arm/Group | Tafamidis
Number analyzed (Participants) | 0

20. Other Pre Specified Outcome: Change From Baseline in Percentage of Left Ventricular Myocardial Mass With Amyloidosis and Left Ventricular Myocardial Mass With Fibrosis/Scar at Month 6 and 12
Description: Cardiac MRI was done to measure percentage of LV myocardial mass with amyloidosis and LV myocardial mass with fibrosis/scar. LV myocardial mass with amyloidosis or fibrosis/scar was calculated from the product of the myocardial volume and specific gravity of heart muscle, in participants with amyloidosis or fibrosis/scar, respectively.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage of LVM
Arm/Group | Tafamidis
Number analyzed (Participants) | 15
Percentage of LVM
  LV Amyloidosis: Baseline (n=15) | 29.069 (11.111)
  LV Amyloidosis: Change at Month 6 (n=14) | -8.200 (14.115)
  LV Amyloidosis: Change at Month 12 (n=9) | -7.017 (13.660)
  LV Fibrosis/Scar: Baseline (n=15) | 36.513 (17.789)
  LV Fibrosis/Scar: Change at Month 6 (n=14) | -10.126 (26.397)
  LV Fibrosis/Scar: Change at Month 12 (n=9) | -8.268 (24.884)

21. Other Pre Specified Outcome: Change From Baseline in 4 Chamber Interatrial Septal Thickness at Month 6 and 12
Description: Cardiac MRI was done to measure interatrial septal thickness in the 4 chamber view.
Time Frame: Baseline, Month 6, Month 12
Population: Data for this measure was not collected due to a change in the planned analysis.
Arm/Group | Tafamidis
Number analyzed (Participants) | 0

22. Other Pre Specified Outcome: Change From Baseline in 4 Chamber Left Atrial Dimension and 4 Chamber Right Atrial Dimension at Month 6 and 12
Description: Cardiac MRI was done to measure the left and right atrial dimensions which have diagnostic and prognostic significance in cardiology, in the 4 chamber view.
Time Frame: Baseline, Month 6, Month 12
Population: Data for this measure was not collected due to a change in the planned analysis.
Arm/Group | Tafamidis
Number analyzed (Participants) | 0

23. Other Pre Specified Outcome: Number of Participants With Atrial Fibrillation/Flutter, Atrial Tachycardia, Non-Sustained Ventricular Tachycardia (NSVT) Beats), Sustained Ventricular Tachycardia (SVT), Sinus Pause at Month 6 and 12
Description: Holter monitor was a machine that recorded the heart rhythms. Holter monitoring abnormalities of atrial fibrillation/flutter (rapid, irregular heart rhythm), atrial tachycardia (rapid cardiac rate), non-sustained ventricular tachycardia (NSVT)<30 beats, sustained ventricular tachycardia (SVT) >=30 beats and sinus pause (transient interruption in the sinus rhythm) were recorded.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Tafamidis
Number analyzed (Participants) | 34
Participants
  Atrial fibrillation/flutter: Baseline (n=33) | 6
  Atrial fibrillation/flutter: Month 6 (n=27) | 9
  Atrial fibrillation/flutter: Month 12 (n=22) | 9
  Atrial tachycardia: Baseline (n=34) | 14
  Atrial tachycardia: Month 6 (n=20) | 0
  Atrial tachycardia: Month 12 (n=17) | 0
  NSVT (<30 beats): Baseline (n=34) | 20
  NSVT (<30 beats): Month 6 (n=13) | 3
  NSVT (<30 beats): Month 12 (n=12) | 5
  SVT (>= 30 beats): Baseline (n=34) | 0
  SVT (>= 30 beats): Month 6 (n=33) | 0
  SVT (>= 30 beats): Month 12 (n=30) | 1
  Sinus pause: Baseline (n=34) | 2
  Sinus pause: Month 6 (n=31) | 4
  Sinus pause: Month 12 (n=28) | 5

24. Other Pre Specified Outcome: 24-Hour Average Heart Rate and Maximium/Minimum Heart Rate
Description: Holter monitor was a machine that recorded the heart rhythms. 24-hour average heart rate and maximium/minimum heart rate was recorded using Holter monitoring.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Tafamidis
Number analyzed (Participants) | 34
beats per minute (bpm)
  24-hour average heart rate: Baseline (n=34) | 74.7 (7.8)
  24-hour average heart rate: Month 6 (n=33) | 73.0 (7.2)
  24-hour average heart rate: Month 12 (n=30) | 76.6 (9.0)
  Maximum Heart Rate: Baseline (n=34) | 111.7 (22.3)
  Maximum Heart Rate: Month 6 (n=33) | 112.3 (17.0)
  Maximum Heart Rate: Month 12 (n=30) | 121.9 (20.4)
  Minimum Heart Rate: Baseline (n=34) | 56.6 (8.0)
  Minimum Heart Rate: Month 6: (n=33) | 53.1 (11.5)
  Minimum Heart Rate Month 12: (n=30) | 55.3 (10.1)

25. Other Pre Specified Outcome: Number of Participants With Complete Heart Block
Description: Complete heart block is the third-degree atrioventricular block in which the impulse generated in the sinoatrial node in the atrium does not propagate to the ventricles.
Time Frame: Baseline, Month 6, Month 12
Population: No summary was prepared for this data as there were no reports of complete heart block.
Arm/Group | Tafamidis
Number analyzed (Participants) | 0

26. Other Pre Specified Outcome: Heart Rate Variability (HRV)- Standard Deviation (SD) Parameters
Description: Holter monitor was a machine that recorded the heart rhythms. HRV time-domain indices were summarized for root-mean-square of successive differences [RMS SD] of the R-R intervals (R-R is the interval between successive Rs in the ECG wave) between normal beats (NN), magid standard deviation (Magid SD) of normal to normal R-R intervals and Kleiger standard deviation of normal to normal R-R intervals (Kleiger SD). The term 'NN' is used in place of 'R-R' when the processed beats are normal beats.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Tafamidis
Number analyzed (Participants) | 33
msec
  HRV- RMS SD: Baseline (n=30) | 75.9 (71.0)
  HRV- RMS SD: Month 6 (n=26) | 88.1 (71.0)
  HRV- RMS SD: Month 12 (n=21) | 91.7 (72.1)
  HRV- Magid SD: Baseline (n=31) | 58.3 (42.1)
  HRV- Magid SD: Month 6 (n=33) | 82.6 (55.5)
  HRV- Magid SD: Month 12 (n=30) | 78.6 (50.1)
  HRV- Kleiger SD: Baseline (n=31) | 100.3 (49.1)
  HRV- Kleiger SD: Month 6 (n=33) | 123.9 (52.8)
  HRV- Kleiger SD: Month 12 (n=30) | 120.3 (48.7)

27. Other Pre Specified Outcome: Heart Rate Variability- Percentage of Successive R-R Intervals With Greater Than 50 Msec Difference Between Normal Beats (pNN50)
Description: Holter monitor was a machine that recorded the heart rhythms. The term 'NN' was used in place of 'R-R' when the processed beats are normal beats. The percentage of successive R-R intervals with greater than 50 msec difference between normal beats was derived by dividing NN50 by the total number of NN intervals (pNN50), where NN50 was the number of interval differences of successive NN intervals greater than 50 msec.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage of intervals
Arm/Group | Tafamidis
Number analyzed (Participants) | 30
Percentage of intervals
  Baseline (n=30) | 19.7 (25.5)
  Month 6 (n=26) | 29.3 (32.7)
  Month 12 (n=21) | 23.6 (27.3)

28. Other Pre Specified Outcome: Number of Participants With Change From Baseline in New York Heart Association (NYHA) Classification at Week 6, Month 3, 6 and 12
Description: NYHA: classified as 'class I' (participants with cardiac disease but without resulting limitations of physical activity), 'class II' (participants with cardiac disease resulting in slight limitation of physical activity), 'class III' (participants with cardiac disease resulting in marked limitation of physical activity), 'class IV' (participants with cardiac disease resulting in inability to carry on any physical activity without discomfort). Participants with change from baseline were classified as 'improved' (positive change), 'no change' or 'worsened' (negative change).
Time Frame: Baseline, Week 6, Month 3, Month 6, Month 12
Population: ITT population included all participants who received at least one dose of study medication. Data at Week 6 was collected but was not summarized due to a change in the planned analysis. Here 'n' signifies those participants who were evaluable for specific timepoints.
Measure: Number; unit: Participants
Arm/Group | Tafamidis
Number analyzed (Participants) | 35
Participants
  Baseline: Class I (n=35) | 5
  Baseline: Class II (n=35) | 28
  Baseline: Class III (n=35) | 2
  Baseline: Class IV (n=35) | 0
  Change at Month 3: improved (n=34) | 5
  Change at Month 3: no change (n=34) | 23
  Change at Month 3: worsened (n=34) | 6
  Change at Month 6: improved (n=34) | 1
  Change at Month 6: no change (n=34) | 27
  Change at Month 6: worsened (n=34) | 6
  Change at Month 12: improved (n=32) | 4
  Change at Month 12: no change (n=32) | 20
  Change at Month 12: worsened (n=32) | 8

29. Other Pre Specified Outcome: Cardiothoracic (CT) Ratio
Description: Cardiothoracic ratio was defined as the transverse diameter of the heart, compared with that of the thoracic cage, used to help determine enlargement of the heart.
Time Frame: Baseline, Month 6, Month 12
Population: ITT population included all participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Tafamidis
Number analyzed (Participants) | 35
Ratio
  Baseline | 55.130 (6.075)
  Month 6 | 56.620 (5.904)
  Month 12 | 57.830 (5.366)

30. Other Pre Specified Outcome: Number of Participants With Increased Interstitial Markings and Pleural Effusions
Description: Chest x-ray was done to record the presence of increased interstitial markings (a large number of interstitial markings was indicative of abnormality in the lung) and pleural effusion, which was defined as accumulation of fluid between the layers of tissue that line the lungs and chest cavity.
Time Frame: Baseline, Month 6, Month 12
Population: Intent to Treat (ITT) population included all participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Tafamidis
Number analyzed (Participants) | 35
Participants
  Increased interstitial markings: Baseline | 11
  Increased interstitial markings: Month 6 | 4
  Increased interstitial markings: Month 12 | 4
  Pleural effusion- right: Baseline | 9
  Pleural effusion- right: Month 6 | 8
  Pleural effusion- right: Month 12 | 6
  Pleural effusion- left: Baseline | 6
  Pleural effusion- left: Month 6 | 5
  Pleural effusion- left: Month 12 | 4
  Pleural effusion- bilateral: Baseline | 6
  Pleural effusion- bilateral: Month 6 | 4
  Pleural effusion- bilateral: Month 12 | 3

31. Other Pre Specified Outcome: Number of Participants With Change in Patient Global Assessment (PtGA) at Month 3, 6 and 12
Description: Participant's overall quality of life was measured by the PtGA. At baseline participants answered to question: "in general, how do you feel today?" - on a 5-point scale from '1' (excellent) to '5' (poor). At each follow-up visit, participant's answered to question: "How do you feel today as compared to when we talked with you at your last clinic visit for this study?" on a 7-point scale- '1' markedly improved, '2' moderately improved, '3' mildly improved, '4' unchanged, '5' mildly worsened, '6' moderately worsened, '7' markedly worsened.
Time Frame: Baseline, Month 3, Month 6, Month 12
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Tafamidis
Number analyzed (Participants) | 34
Participants
  Excellent: Baseline (n=33) | 5
  Very good: Baseline (n=33) | 14
  Good: Baseline (n=33) | 12
  Fair: Baseline (n=33) | 2
  Poor: Baseline (n=33) | 0
  Markedly improved: Month 3 (n=34) | 2
  Moderately improved: Month 3 (n=34) | 7
  Mildly improved: Month 3 (n=34) | 6
  Unchanged: Month 3 (n=34) | 15
  Mildly worsened: Month 3 (n=34) | 2
  Moderately worsened: Month 3 (n=34) | 2
  Markedly worsened: Month 3 (n=34) | 0
  Markedly improved: Month 6 (n=34) | 3
  Moderately improved: Month 6 (n=34) | 4
  Mildly improved: Month 6 (n=34) | 3
  Unchanged: Month 6 (n=34) | 16
  Mildly worsened: Month 6 (n=34) | 8
  Moderately worsened: Month 6 (n=34) | 0
  Markedly worsened: Month 6 (n=34) | 0
  Markedly improved: Month 12 (n=32) | 0
  Moderately improved: Month 12 (n=32) | 5
  Mildly improved: Month 12 (n=32) | 3
  Unchanged: Month 12 (n=32) | 16
  Mildly worsened: Month 12 (n=32) | 4
  Moderately worsened: Month 12 (n=32) | 3
  Markedly worsened: Month 12 (n=32) | 1

32. Other Pre Specified Outcome: Change From Baseline in Kansas City Cardiomyopathy Questionnaire (KCCQ) Score at Month 3, 6 and 12
Description: KCCQ was a 23-item heart failure specific questionnaire quantified in to following 10 summary scores: physical limitation, symptom frequency, symptom severity, and symptom stability, total symptoms, quality of life, social interference, self-efficacy, overall summary and clinical summary. Total score ranged from 0 to 100, where higher scores indicated better functioning, fewer symptoms, and better disease specific quality of life. Summary scores were scaled to range from 0 to 100, with higher scores representing greater disability.
Time Frame: Baseline, Month 3, Month 6, Month 12
Population: ITT population included all participants who received at least one dose of study medication. Here 'n' signifies those participants who were evaluable for specific timepoints.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tafamidis
Number analyzed (Participants) | 35
Units on a scale
  Physical limitations: Baseline (n=35) | 72.9 (20.8)
  Physical limitations: Change at Month 3 (n=33) | -2.7 (15.0)
  Physical limitations: Change at Month 6 (n=34) | -0.4 (13.6)
  Physical limitations: Change at Month 12 (n=31) | -8.1 (18.8)
  Symptom stability: Baseline (n=35) | 55.7 (13.7)
  Symptom stability: Change at Month 3 (n=34) | 3.7 (27.6)
  Symptom stability: Change at Month 6 (n=34) | -5.9 (25.4)
  Symptom stability: Change at Month 12 (n=31) | 0.0 (22.4)
  Symptom frequency: Baseline (n=35) | 73.8 (22.2)
  Symptom frequency: Change at Month 3 (n=34) | -1.8 (18.5)
  Symptom frequency: Change at Month 6 (n=34) | -2.5 (15.9)
  Symptom frequency: Change at Month 12 (n=31) | -6.0 (18.2)
  Symptom burden: Baseline (n=35) | 76.9 (18.1)
  Symptom burden: Change at Month 3 (n=34) | -4.0 (18.3)
  Symptom burden: Change at Month 6 (n=34) | -4.7 (15.2)
  Symptom burden: Change at Month 12 (n=31) | -8.6 (19.2)
  Total symptom: Baseline (n=35) | 75.4 (19.2)
  Total symptom: Change at Month 3 (n=34) | -2.9 (16.9)
  Total symptom: Change at Month 6 (n=34) | -3.6 (14.3)
  Total symptom: Change at Month 12 (n=31) | -7.3 (18.2)
  Self-efficacy: Baseline (n=35) | 85.7 (19.0)
  Self-efficacy: Change at Month 3 (n=33) | 1.9 (14.7)
  Self-efficacy: Change at Month 6 (n=34) | 1.1 (13.5)
  Self-efficacy: Change at Month 12 (n=31) | 1.6 (16.7)
  Quality of life: Baseline (n=35) | 66.9 (19.2)
  Quality of life: Change at Month 3 (n=34) | 1.0 (18.2)
  Quality of life: Change at Month 6 (n=34) | -0.2 (14.4)
  Quality of life: Change at Month 12 (n=31) | -4.0 (20.4)
  Social limitation: Baseline (n=33) | 69.3 (25.4)
  Social limitation: Change at Month 3 (n=30) | -0.6 (19.6)
  Social limitation: Change at Month 6 (n=31) | -2.4 (22.6)
  Social limitation: Change at Month 12 (n=27) | -9.2 (25.2)
  Overall summary: Baseline (n=35) | 71.4 (18.8)
  Overall summary: Change at Month 3 (n=34) | -0.8 (14.9)
  Overall summary: Change at Month 6 (n=34) | -1.5 (12.4)
  Overall summary: Change at Month 12 (n=31) | -6.9 (18.0)
  Clinical summary: Baseline (n=35) | 74.1 (18.9)
  Clinical summary: Change at Month 3 (n=34) | -2.0 (15.9)
  Clinical summary: Change at Month 6 (n=34) | -2.0 (11.9)
  Clinical summary: Change at Month 12 (n=31) | -7.7 (17.9)

33. Other Pre Specified Outcome: Change From Baseline in the Short Form 36 (SF-36) at Month 3, 6 and 12
Description: SF-36 was standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. Scores for the 8 domains range from 0-100, where higher scores were better (100=highest level of functioning) and reported as 2 summary scores; Mental Component Score (MCS) and Physical Component Score (PCS). The score for a section was an average of the individual question scores, which were scaled 0-100, where higher scores were better.
Time Frame: Baseline, Month 3, Month 6, Month 12
Population: ITT population included all participants who received at least one dose of study medication. Here 'n' signifies those participants who were evaluable for specific timepoints. Data was collected at Month 3 but not statistically summarized as planned.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tafamidis
Number analyzed (Participants) | 35
Units on a scale
  PCS: Baseline (n=33) | 41.0 (9.69)
  PCS: Change at Month 6 (n=32) | -1.4 (5.87)
  PCS: Change at Month 12 (n=29) | -2.4 (7.58)
  MCS: Baseline (n=33) | 52.7 (9.51)
  MCS: Change at Month 6 (n=32) | 0.3 (8.40)
  MCS: Change at Month 12 (n=29) | -2.0 (9.56)
  Physical functioning: Baseline (n=34) | 37.7 (11.28)
  Physical functioning: Change at Month 6 (n=33) | -0.7 (6.89)
  Physical functioning: Change at Month 12 (n=29) | -2.0 (7.34)
  Role-physical: Baseline (n=35) | 42.3 (10.84)
  Role-physical: Change at Month 6 (n=34) | -1.4 (7.12)
  Role-physical: Change at Month 12 (n=30) | -3.5 (9.29)
  Bodily pain: Baseline (n=35) | 53.2 (9.57)
  Bodily pain: Change at Month 6 (n=34) | -4.0 (8.74)
  Bodily pain: Change at Month 12 (n=30) | -3.2 (11.81)
  General health: Baseline (n=35) | 41.5 (9.33)
  General health: Change at Month 6 (n=34) | 0.7 (9.23)
  General health: Change at Month 12 (n=30) | -1.6 (8.44)
  Vitality: Baseline (n=34) | 50.6 (8.11)
  Vitality: Change at Month 6 (n=33) | -0.1 (6.83)
  Vitality: Change at Month 12 (n=30) | -2.2 (7.83)
  Social functioning: Baseline (n=35) | 48.4 (9.84)
  Social functioning: Change at Month 6 (n=34) | -2.9 (9.23)
  Social functioning: Change at Month 12 (n=30) | -3.6 (11.40)
  Role-emotional: Baseline (n=35) | 45.2 (11.71)
  Role-emotional: Change at Month 6 (n=34) | 0.6 (12.26)
  Role-emotional: Change at Month 12 (n=30) | -3.0 (12.53)
  Mental health: Baseline (n=34) | 53.3 (8.50)
  Mental health: Change at Month 6 (n=33) | 0.3 (5.01)
  Mental health: Change at Month 12 (n=30) | -1.1 (7.50)

34. Other Pre Specified Outcome: Change From Baseline in Troponin I and Troponin T at Week 2, 6, Month 3, 6 and 12
Description: Troponin I and troponin T were the cardiac markers. Troponin I and troponin T were part of the troponin complex, where troponin I was bound to actin in thin myofilaments and troponin T was bound to tropomyosin. Higher level of these markers was indicative of heart damage.
Time Frame: Baseline, Week 2, Week 6, Month 3, Month 6, Month 12
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Tafamidis
Number analyzed (Participants) | 35
nanogram/milliliter (ng/mL)
  Troponin I: Baseline (n=33) | 0.135 (0.080)
  Troponin I: Change at Week 2 (n=35) | 0.003 (0.060)
  Troponin I: Change at Week 6 (n=35) | -0.000 (0.055)
  Troponin I: Change at Month 3 (n=34) | 0.008 (0.057)
  Troponin I: Change at Month 6 (n=34) | -0.016 (0.051)
  Troponin I: Change at Month 12 (n=32) | 0.016 (0.064)
  Troponin T: Baseline (n=33) | 0.044 (0.037)
  Troponin T: Change at Week 2 (n=35) | 0.001 (0.025)
  Troponin T: Change at Week 6 (n=35) | 0.006 (0.020)
  Troponin T: Change at Month 3 (n=34) | 0.008 (0.021)
  Troponin T: Change at Month 6 (n=33) | 0.002 (0.020)
  Troponin T: Change at Month 12 (n=32) | 0.012 (0.023)

35. Other Pre Specified Outcome: Change From Baseline in N-Terminal Prohormone Brain Natriuretic Peptide(NT-proBNP) Levels at Week 2, 6, Month 3, 6 and 12
Description: NT-proBNP was a cardiac marker which had the prognostic value for participants with heart failure or left ventricular dysfunction. Higher level of the marker was indicative of heart damage.
Time Frame: Baseline, Week 2, Week 6, Month 3, Month 6, Month 12
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: picogram/mL (pg/mL)
Arm/Group | Tafamidis
Number analyzed (Participants) | 35
picogram/mL (pg/mL)
  Baseline (n=33) | 4934.2 (4324.9)
  Change at Week 2 (n=35) | -1.6 (1349.1)
  Change at Week 6 (n=35) | 295.0 (1632.0)
  Change at Month 3 (n=34) | 102.8 (1998.0)
  Change at Month 6 (n=33) | 111.6 (2032.4)
  Change at Month 12 (n=31) | 958.2 (3178.0)

36. Other Pre Specified Outcome: Change From Baseline in 6-Minute Walk Test (6MWT) at Month 3, 6 and 12
Description: 6MWT was used to assess the distance that a participant could walk in 6 minutes. Participants were asked to perform the test at a pace that was comfortable to them, with as many breaks as they needed. Continuous pulse oximetry was conducted during the test for safety.. The distance walked in 6 minutes was categorized as: Level 1: <300 meter, Level 2: 300-374.9 meter, Level 3: 375-449.9 meter, Level 4: >=450 meter.
Time Frame: Baseline, Month 3, Month 6, Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Tafamidis
Number analyzed (Participants) | 34
meters
  Distance walked: Baseline (n=34) | 354.5 (126.0)
  Distance walked: Change at Month 3 (n=31) | -4.6 (63.1)
  Distance walked: Change at Month 6 (n=33) | 3.9 (58.2)
  Distance walked: Change at Month 12 (n=28) | -11.2 (76.4)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Tafamidis
Serious Adverse Events (participants affected / at risk) | 15/35
Other Adverse Events (participants affected / at risk) | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tafamidis (N=35)
Cardiac failure congestive (Cardiac disorders) | 9
Atrial fibrillation (Cardiac disorders) | 3
Cardiac failure (Cardiac disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Amyloidosis (Immune system disorders) | 1
Cellulitis (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 3
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Syncope (Nervous system disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 1
Coordination abnormal (Nervous system disorders) | 1
Haemorrhagic stroke (Nervous system disorders) | 1
Metabolic encephalopathy (Nervous system disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Haemorrhage (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tafamidis (N=35)
Anaemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 4
Cardiac failure congestive (Cardiac disorders) | 3
Cardiac failure (Cardiac disorders) | 2
Atrial tachycardia (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Bundle branch block right (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus arrhythmia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Colour blindness (Congenital, familial and genetic disorders) | 1
Corneal disorder (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 3
Dry mouth (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Faecal incontinence (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 8
Oedema peripheral (General disorders) | 6
Asthenia (General disorders) | 3
Oedema (General disorders) | 3
Thirst (General disorders) | 3
Catheter related complication (General disorders) | 1
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Hernia (General disorders) | 1
Hot flush (General disorders) | 1
Localised oedema (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Hepatomegaly (Hepatobiliary disorders) | 4
Seasonal allergy (Immune system disorders) | 3
Upper respiratory tract infection (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 3
Influenza (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Nail infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Excoriation (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 2
Joint injury (Injury, poisoning and procedural complications) | 2
Skin laceration (Injury, poisoning and procedural complications) | 2
Joint sprain (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 1
Tooth injury (Injury, poisoning and procedural complications) | 1
Weight decreased (Investigations) | 6
Work increased (Investigations) | 5
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood cholesterol increased (Investigations) | 2
Blood thyroid stimulating hormone increased (Investigations) | 2
Aspiration pleural cavity (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood pressure decreased (Investigations) | 1
Blood thyroid stimulating hormone decreased (Investigations) | 1
Blood urine present (Investigations) | 1
Blood natriuretic peptide increased (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Heart rate increased (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Urine output increased (Investigations) | 1
Venous pressure jugular increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 2
Fluid overload (Metabolism and nutrition disorders) | 2
Gout (Metabolism and nutrition disorders) | 2
Fluid retention (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypochloraemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Finger deformity (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lentigo (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 7
Dizziness postural (Nervous system disorders) | 6
Balance disorder (Nervous system disorders) | 5
Aguesia (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 2
Amnesia (Nervous system disorders) | 1
Disturbance in attention (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Neuropathy (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Restless legs syndrome (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 3
Confusional state (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 1
Nervousness (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Nipple pain (Reproductive system and breast disorders) | 2
Gynaecomastia (Reproductive system and breast disorders) | 1
Scrotal oedema (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 3
Blister (Skin and subcutaneous tissue disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Foot operation (Surgical and medical procedures) | 1
Implantable defibrillator insertion (Surgical and medical procedures) | 1
Mole excision (Surgical and medical procedures) | 1
Tooth extraction (Surgical and medical procedures) | 1
Hypotension (Vascular disorders) | 1
Varicose vein (Vascular disorders) | 1
Bundle branch block (Cardiac disorders) | 1

LIMITATIONS AND CAVEATS:
Results for Holter monitoring parameters, increased interstitial markings, pleural effusions, PtGA and cardiothoracic ratio are presented as absolute values at specified time points and not as change from baseline as planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.